CLINICAL TRIAL: NCT06975358
Title: Impact of Alveolar Decortication Combined With CGF Injection on Acceleration of Maxillary Canine Retraction-A Randomized Clinical Trial
Brief Title: Accelerated Orthodontics With Alveolar Decortication Plus CGF Injection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Safa Basiouny Alawy (Other)
Responsible Party: Sponsor-Investigator, Safa Basiouny Alawy, Lecturer of Orthodontics, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #R-OS-12-24-3158
Record Dates: First submitted 2025-05-08; First posted 2025-05-16 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Accelerate Tooth Movement
MeSH Terms: interventions — Acceleration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alveolar decortication plus CGF (Experimental): Alveolar decortication followed by submucosal CGF injection (70 units) disto-buccal and disto-palatal to the maxillary canine will be randomly assigned to one side of the maxillary arch (experimental) while the other side serve as (control) receiving orthodontic treatment without any additional intervention
  Interventions: Procedure: Alveolar decortication plus CGF injection
- Control (Active Comparator): the other side of the maxillary arch will receive the usual orthodontic treatment without any additional intervention
  Interventions: Procedure: canine retraction without acceleration

INTERVENTIONS:
Procedure: Alveolar decortication plus CGF injection — Experimental sides will receive CGF injection (70 units) disto-buccal and disto-palatal to the maxillary canine after performing decortication. After administration of local anesthesia, two-line flap will be performed from the mesial surface of the maxillary second premolar to the distal surface of the maxillary canine Mucoperiosteal flap will be reflected in the buccal side. Two millimeters of marginal crestal bone will be held intact and using a high-speed drill and a round carbide bur (1mm diameter) under copious saline irrigation, the cortical wall will be penetrated to reach marrow spaces. Multiple perforations (10 holes for standardization) in the cortical bone will be created. The surgical site will then rinsed, and the flap will be repositioned and sutured.
  Arms: Alveolar decortication plus CGF
Procedure: canine retraction without acceleration — in the control side, the maxillary canine will be retracted without any acceleration procedure
  Arms: Control

SUMMARY:
The aim of the present study is to evaluate alveolar bone decortication combined with CGF Injection on tooth movement acceleration

ELIGIBILITY:
Inclusion Criteria:

1. Age of the patients ranged from 16: 22 years old.
2. Malocclusion that requires extraction of the maxillary first premolar and canine retraction (e.g. class I bimaxillary dentoalveolar protrusion and class II div 1 malocclusion).
3. Maximum anchorage needed for the maxillary arch as a part of the orthodontic treatment plan.
4. Good oral hygiene and periodontal condition.

Exclusion Criteria:

1. Medically compromised patients.
2. Severe crowding in the maxillary arch.
3. Chronic intake of NSAIDs or any medication that interfere with OTM.
4. Previous orthodontic treatment.

Ages: 16 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
rate of canine retraction | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, Tanta, Egypt